CLINICAL TRIAL: NCT06857526
Title: The Relationship of Hand Sensory and Strength Assessments with Functionality and Kinesiophobia in Individuals with Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Esra, physiotherapy and rehabilitation, Firat University
Other Study IDs: FiratU-FTR
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Disease
Keywords: hand force assessment; hand sensory evaluation; romatoid artrit
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Romatoid artrit: Patient diagnosed with RA according to the American College of Rheumatology (ACR) criteria

SUMMARY:
Rheumatoid arthritis (RA) is a systemic inflammatory disease that can involve all tissues with synovium. The wrist and hand, which are of great importance in our daily activities, are involved early and specifically because they are rich in synovium, which is the target tissue in RA.In many patients with rheumatoid arthritis, hand and wrist involvement is seen from the early stages of the disease. Pain, stiffness and swelling in the joint are accompanied by decreased range of motion and muscle strength.Hand functions have a very important place due to the fact that the hand must be used in countless daily life activities.Kinesiophobia is defined as a state of fear and avoidance of activity and physical movement caused by painful injury and sensitivity to repeated injury.The aim of this study was to investigate the relationship between hand sensory and strength assessment, functionality and kinesiophobia in individuals with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic inflammatory disease that can involve all tissues with synovium. The wrist and hand, which are of great importance in our daily activities, are involved early and specifically because they are rich in synovium, which is the target tissue in RA.In many patients with rheumatoid arthritis, hand and wrist involvement is seen from the early stages of the disease. Pain, stiffness and swelling in the joint are accompanied by decreased range of motion and muscle strength.Hand functions have a very important place due to the fact that the hand must be used in countless daily life activities.Kinesiophobia is defined as a state of fear and avoidance of activity and physical movement caused by painful injury and sensitivity to repeated injury.The aim of this study was to investigate the relationship between hand sensory and strength assessment, functionality and kinesiophobia in individuals with rheumatoid arthritis.Thirty patients who were followed up in the Rheumatology outpatient clinic of Fırat University Hospital and diagnosed with RA according to the American College of Rheumatology (ACR) criteria will be included. SPSS program will be used in statistical analysis. Descriptive statistics will be used for the demographic characteristics of the groups. Qualitative variables will be defined by number and quantitative variables will be defined by mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18-65 years of age
* Patients whose medical treatment has been stable for the last 3 months

Exclusion Criteria:

* Patients who have undergone surgery on the hand and wrist
* Patients with prosthesis
* Patients with neurological or orthopedic diseases
* Patients with another accompanying rheumatic disease
* Patients with malignancy
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
hand sensory evaluation | 15 minutes
  Semmes-Weinstein Monofilaments will be used to measure light touch sensation.This test is performed with the patient's head turned to the other side.The monofilaments are held perpendicular to the skin and pressed against the skin until there is a slight curvature. The test is performed 3 times for monofilaments from 1.65 to 4.08 to obtain a stimulus response. 1 time for monofilaments from 4.17 to 6.65. If the patient hidded this monofilament, the test is finished. If the patient does not respond to the stimulus, the test is switched to the thicker filament and continued until the patient feels it.

IPD SHARING:
Plan to Share IPD: Undecided